CLINICAL TRIAL: NCT01630135
Title: Study FFR116364, a Double-blind, Placebo-controlled Study of GW685698X in Paediatric Subjects With Perennial Allergic Rhinitis
Brief Title: Study FFR116364, a Placebo-controlled Study of GW685698X in Paediatric Subjects With Perennial Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 116364
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Results first posted 2013-05-01 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-11

CONDITIONS: Rhinitis, Allergic, Perennial
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — fluticasone furoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- GW685698X (Experimental): GW685698X 55mcg/day
  Interventions: Drug: Fluticasone furoate
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluticasone furoate — 55 mcg/day, intranasal, 2 weeks
  Arms: GW685698X
Drug: Placebo — Placebo, intranasal, 2 weeks
  Arms: Placebo

SUMMARY:
Efficacy and safety of GW685698X (55 µg/day, q.d.) nasal spray over a period of 2 weeks in Japanese paediatric subjects ages 6 to < 15 years with perennial allergic rhinitis will be evaluated compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* 6 to <15 years of age, male or eligible female (females of childbearing potential must commit to consistent and correct use of an acceptable method of birth control), outpatient
* Diagnosis of perennial allergic rhinitis: A positive test response to house dust and/or dust mites on serum antigen-specific IgE antibody test at Visit 1. One year or more clinical history of perennial allergic rhinitis. A positive test result on nasal eosinophil count at Visit 1/1A.
* Either subject's parent/guardian who signed ICF or subject is able to complete assessments on the patient diary through the study.
* ALT < 2xULN; alkaline phosphatase and bilirubin <= 1.5xULN
* Average of 3TNSS is >= 4.0 in the last consecutive 4 days prior to Visit 2.
* Completion of the patient diary on >= 3 days of the last consecutive 4 days prior to Visit 2

Exclusion Criteria:

* Has a seasonal pollen as an allergen
* A nose disorder that could affect the assessment of the study medication or eye or nose surgery (within 3 months prior to Visit 1)
* Bacterial or viral infection of upper respiratory tract or eye
* Concurrent disease/abnormalities: Clinically significant uncontrolled disease
* Known hypersensitivity to corticosteroids or any excipients in the investigational product
* Has recent participation in a study and/or exposure to an investigational study drug within 3 months prior to Visit 1
* Use of the following medication and/or its combination drug within the specified time:

Anti-IgE (Within 6 months prior to Visit 1), Immunosuppressive medications or Systemic corticosteroids (Within 8 weeks prior to Visit 1), Topical corticosteroids (Within 4 weeks prior to Visit 1), Immunotherapy or nonspecific allassotherapy which was initiated, discontinued or changed its dose within 4 weeks prior to Visit 1

* Affiliation with Investigator's Site: Relative or employee
* History of alcohol or drug abuse, children in care or in the opinion of the investigator (sub-investigator), inappropriate to be enrolled in the study.
* Average of 3TNSS is >= 8.0 in the last consecutive 4 days prior to Visit 2.
* Bacterial or viral infection of upper respiratory tract or eye during the screening period.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 261 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- Japan (6):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Gifu
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 116364 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116364 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116364 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116364 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Fluticasone Furoate 55 µg Per Day: Fluticasone furoate nasal spray (55 micrograms [µg] per day) was administered as one spray into each nostril (27.5 μg per spray) once daily in the morning for 2 weeks.
- Placebo: Matching placebo nasal spray was administered as one spray into each nostril once daily in the morning for 2 weeks.
Period: Overall Study
Arm/Group | Fluticasone Furoate 55 µg Per Day | Placebo
Started | 131 | 130
Completed | 131 | 128
Not Completed | 0 | 2
Not completed — Protocol-defined Stopping Criteria Met | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluticasone Furoate 55 µg Per Day | Placebo | Total
Number analyzed (Participants) | 131 | 130 | 261
Age, Continuous [Mean (Standard Deviation); unit: Years] | 10.0 (2.32) | 10.1 (2.22) | 10.1 (2.26)
Gender [Count of Participants; unit: Participants]
  Female | 46 | 51 | 97
  Male | 85 | 79 | 164
Race/Ethnicity, Customized [Number; unit: participants]
  Asian - Japanese Heritage | 131 | 130 | 261

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the 3 Total Nasal Symptom Score (3TNSS) Over the Entire Treatment Period
Description: The 3TNSS is the sum of the 3 individual symptom scores for sneezing, rhinorrhea, and nasal congestion. Each symptom is scored on a scale from 0 to 3; the range of sums for the 3TNSS is 0 to 9. The symptoms were evaluated using a scale of 0, 1, 2, or 3; a larger score indicates more severe symptoms. The participant's parent/guardian who signed the informed consent form (ICF) or the participant themself scored nasal symptoms every day during the screening period and the treatment period. The Baseline value is defined as the average 3TNSS over the last 4 consecutive days prior to Visit 2 (start of the treatment period). For the entire assessment period, a mean score for each participant was calculated using available diary data from the assessment periods, taking the average of non-missing data during the period. Change from Baseline was calculated as the mean score for the entire treatment period minus the score at Baseline.
Time Frame: Baseline through the entire treatment period (2 weeks)
Population: Full Analysis Set (FAS): all participants meeting the primary criteria for enrollment, without any major good clinical practice (GCP) deviation, who received at least one dose of the assigned treatment and had diary assessment for 3TNSS after receiving a dose of study medication
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Fluticasone Furoate 55 µg Per Day | Placebo
Number analyzed (Participants) | 131 | 130
Scores on a scale | -1.98 (0.12) | -0.89 (0.12)
Statistical Analysis 1: Comparison: Fluticasone Furoate 55 µg Per Day vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -1.089, 95% CI 2-sided [-1.41 to -0.76] — The analysis was based on an analysis of covariance (ANCOVA) with a model adjusting for Treatment, Baseline, Age, and Sex

2. Secondary Outcome: Mean Change From Baseline in 3TNSS at Week 1 and Week 2
Description: The 3TNSS is the sum of the 3 individual symptom scores for sneezing, rhinorrhea, and nasal congestion. Each symptom is scored on a scale from 0 to 3; the range of sums for the 3TNSS is 0 to 9. The symptoms were evaluated using a scale of 0, 1, 2, or 3; a larger score indicates more severe symptoms. The participant's parent/guardian who signed the ICF or the participant themself scored nasal symptoms every day during the screening period and the treatment period. The Baseline value is defined as the average 3TNSS over the last 4 consecutive days prior to Visit 2 (start of the treatment period). For Week 1 and Week 2, a mean score for each participant was calculated using available diary data from the assessment periods, taking the average of non-missing data during the period. Change from Baseline was calculated as the mean score at Week 1 and Week 2 minus the score at Baseline.
Time Frame: Baseline; Week 1 and Week 2
Population: FAS. Change from Baseline was analyzed for only those participants who were available for assessment at both Baseline and the indicated assessment period. The analysis was based on ANCOVA with a model adjusting for Treatment, Baseline, Age, and Sex.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Fluticasone Furoate 55 µg Per Day | Placebo
Number analyzed (Participants) | 131 | 130
Scores on a scale
  Week 1, n=131, 130 | -1.60 (0.12) | -0.70 (0.12)
  Week 2, n=131, 128 | -2.38 (0.13) | -1.10 (0.13)

3. Secondary Outcome: Mean Percent Change From Baseline in 3TNSS Over the Entire Treatment Period, at Week 1, and at Week 2
Description: The 3TNSS is the sum of the 3 individual symptom scores for sneezing, rhinorrhea, and nasal congestion. Each symptom is scored on a scale from 0 to 3; the range of sums for the 3TNSS is 0 to 9. The symptoms were evaluated using a scale of 0, 1, 2, or 3; a larger score indicates more severe symptoms. The participant's parent/guardian who signed the ICF or the participant themself scored nasal symptoms every day during the screening period and the treatment period. The Baseline value is defined as the average 3TNSS over the last 4 consecutive days prior to Visit 2 (start of the treatment period). For the entire treatment period (Weeks 1 and 2), Week 1, and Week 2, a mean score for each participant was calculated using available diary data from the assessment periods, taking the average of non-missing data during the period. Percent change from Baseline=(mean score at the post-Baseline assessment minus the score at Baseline) divided by the Baseline value * 100.
Time Frame: Baseline through the entire treatment period (2 weeks), Week 1, and Week 2
Population: FAS. Only those participants who were available for assessment at both Baseline and the indicated assessment period were analyzed. Participants were analyzed for the entire treatment period if they had an assessment on any day during Week 1 and Week 2. The analysis was based on an ANCOVA with a model adjusting for Treatment, Baseline, Age, and Sex.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Fluticasone Furoate 55 µg Per Day | Placebo
Number analyzed (Participants) | 131 | 130
Percent change
  Entire treatment period, n=131, 130 | -39.76 (2.38) | -17.74 (2.36)
  Week 1, n=131, 130 | -31.96 (2.46) | -13.89 (2.44)
  Week 2, n=131, 128 | -47.89 (2.70) | -21.95 (2.70)

4. Secondary Outcome: Mean Change From Baseline in 3TNSS at the Indicated Days
Description: The 3TNSS is the sum of the 3 individual symptom scores for sneezing, rhinorrhea, and nasal congestion. Each symptom is scored on a scale from 0 to 3; the range of sums for the 3TNSS is 0 to 9. The symptoms were evaluated using a scale of 0, 1, 2, or 3; a larger score indicates more severe symptoms. The participant's parent/guardian who signed the ICF or the participant themself scored nasal symptoms every day during the screening period and the treatment period. The Baseline value is defined as the average 3TNSS over the last 4 consecutive days prior to Visit 2 (start of the treatment period). Change from Baseline was calculated as the mean score at the indicated day minus the score at Baseline.
Time Frame: Baseline; Days 1 through 14
Population: FAS. Change from Baseline was analyzed for only those participants who were available for assessment at both Baseline and the indicated study day (Days 1 through 14). The analysis was based on an ANCOVA with a model adjusting for Treatment, Baseline, Age, and Sex.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Fluticasone Furoate 55 µg Per Day | Placebo
Number analyzed (Participants) | 131 | 130
Scores on a scale
  Day 1, n=130, 130 | -0.71 (0.13) | -0.52 (0.12)
  Day 2, n=131, 130 | -1.33 (0.14) | -0.41 (0.14)
  Day 3, n=131, 130 | -1.53 (0.15) | -0.61 (0.15)
  Day 4, n=131, 130 | -1.69 (0.15) | -0.77 (0.15)
  Day 5, n=131, 130 | -1.89 (0.16) | -0.77 (0.16)
  Day 6, n=131, 130 | -1.95 (0.16) | -0.97 (0.16)
  Day 7, n=131, 130 | -2.05 (0.16) | -0.87 (0.16)
  Day 8, n=131, 128 | -2.14 (0.16) | -1.05 (0.16)
  Day 9, n=131, 128 | -2.29 (0.16) | -1.07 (0.16)
  Day 10, n=131, 128 | -2.32 (0.16) | -1.01 (0.16)
  Day 11, n=131, 128 | -2.36 (0.16) | -1.19 (0.16)
  Day 12, n=131, 128 | -2.54 (0.15) | -1.21 (0.15)
  Day 13, n=122, 123 | -2.47 (0.16) | -1.20 (0.16)
  Day 14, n=105, 115 | -2.65 (0.17) | -0.93 (0.16)

5. Secondary Outcome: Mean Change From Baseline in the 4 Total Nasal Symptom Score (4TNSS) Over the Entire Treatment Period, at Week 1, and at Week 2
Description: The 4TNSS is the sum of the 4 individual symptom scores for sneezing, rhinorrhea, nasal congestion, and nasal itching. Each symptom is scored on a scale from 0 to 3; the range of sums for the 4TNSS is 0 to 12. The symptoms were evaluated using a scale of 0, 1, 2, or 3; a larger score indicates more severe symptoms. The participant's parent/guardian who signed the ICF or the participant themself scored nasal symptoms every day during the screening period and the treatment period. The Baseline value is defined as the average of the 4TNSS in the last 4 consecutive days prior to Visit 2 (start of the treatment period). A mean score for each participant was calculated using available diary data from the assessment periods, taking the average of non-missing data during the period. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline through the entire treatment period (2 weeks), Week 1, and Week 2
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Fluticasone Furoate 55 µg Per Day | Placebo
Number analyzed (Participants) | 131 | 130
Scores on a scale
  Entire Treatment Period, n=131, 130 | -2.40 (0.15) | -1.01 (0.15)
  Week 1, n=131, 130 | -1.94 (0.15) | -0.74 (0.15)
  Week 2, n= 131, 128 | -2.89 (0.16) | -1.29 (0.16)

6. Secondary Outcome: Mean Percent Change From Baseline in the 4TNSS Over the Entire Treatment Period, at Week 1, and at Week 2
Description: The 4TNSS is the sum of the 4 individual symptom scores for sneezing, rhinorrhea, nasal congestion, and nasal itching. Each symptom is scored on a scale from 0 to 3; the range of sums for the 4TNSS is 0 to 12. The symptoms were evaluated using a scale of 0, 1, 2, or 3; a larger score indicates more severe symptoms. The participant's parent/guardian who signed the ICF or the participant themself scored nasal symptoms every day during the screening period and the treatment period. The Baseline value is defined as the average 4TNSS over the last 4 consecutive days prior to Visit 2 (start of the treatment period). For the entire treatment period (Weeks 1 and 2), Week 1, and Week 2, a mean score for each participant was calculated using available diary data from the assessment periods, taking the average of non-missing data during the period. Percent change from Baseline=(mean score at the post-Baseline assessment minus the score at Baseline) divided by the Baseline value * 100.
Time Frame: Baseline through the entire treatment period (2 weeks), Week 1, and Week 2
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Fluticasone Furoate 55 µg Per Day | Placebo
Number analyzed (Participants) | 131 | 130
Percent change
  Entire Treatment Period, n=131, 130 | -40.42 (2.46) | -16.09 (2.44)
  Week 1, n=131, 130 | -32.55 (2.54) | -11.54 (2.52)
  Week 2, n= 131, 128 | -48.58 (2.78) | -20.92 (2.78)

7. Secondary Outcome: Mean Change From Baseline in Rhinorrhea, Nasal Congestion, Sneezing, and Nasal Itching Over the Entire Treatment Period (ETP), at Week 1, and at Week 2
Description: Four individual symptoms (sneezing, rhinorrhea, nasal congestion, and nasal itching) were scored on a scale from 0 to 3 using a scale of 0, 1, 2, or 3; a larger score indicates more severe symptoms. The participant's parent/guardian who signed the ICF or the participant themself scored nasal symptoms every day during the screening period and the treatment period. The Baseline value is defined as the average of the symptom scores in the last 4 consecutive days prior to Visit 2 (start of the treatment period). A mean score for each participant was calculated using available diary data from the assessment periods, taking the average of non-missing data during the period. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline through the entire treatment period (2 weeks), Week 1, and Week 2
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Fluticasone Furoate 55 µg Per Day | Placebo
Number analyzed (Participants) | 131 | 130
Scores on a scale
  Rhinorrhea, ETP, n=131, 130 | -0.69 (0.05) | -0.31 (0.05)
  Rhinorrhea, Week 1, n=131, 130 | -0.55 (0.05) | -0.23 (0.05)
  Rhinorrhea, Week 2, n=131, 128 | -0.85 (0.06) | -0.40 (0.06)
  Nasal congestion, ETP, n=131, 130 | -0.70 (0.05) | -0.36 (0.05)
  Nasal congestion, Week 1, n=131, 130 | -0.56 (0.05) | -0.29 (0.05)
  Nasal congestion, Week 2, n=131, 128 | -0.84 (0.05) | -0.43 (0.05)
  Sneezing, ETP, n=131, 130 | -0.60 (0.04) | -0.21 (0.04)
  Sneezing, Week 1, n=131, 130 | -0.50 (0.04) | -0.16 (0.04)
  Sneezing, Week 2, n= 131, 128 | -0.71 (0.05) | -0.27 (0.05)
  Nasal itching, ETP, n=131, 130 | -0.41 (0.04) | -0.12 (0.04)
  Nasal itching, Week 1, n=131, 130 | -0.33 (0.05) | -0.04 (0.05)
  Nasal itching, Week 2, n= 131, 128 | -0.49 (0.05) | -0.19 (0.05)

8. Secondary Outcome: Mean Change From Baseline in the Total Ocular Symptom Score (TOSS) Over the Entire Treatment Period, at Week 1, and at Week 2
Description: Symptoms of eye itching, tearing, and redness were scored by the participant's parent/guardian who signed the ICF or the participant themself using a scale of 0, 1, 2, or 3 (a larger score indicates more severe symptoms) and were recorded in the participant's diary. The TOSS is the sum of all three symtpom scores and ranges from 0 to 9. The mean of the Baseline period is defined as the mean score of 4 consecutive days prior to Visit 2 (start of the treatment period). The mean of each assessment period is defined as the mean score of the entire treatment period (Weeks 1 and 2), Week 1, and Week 2. For each assessment period, a mean score for each participant was calculated using available diary data from the assessment periods, taking the average of non-missing data during the period. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline through the entire treatment period (2 weeks), Week 1, and Week 2
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Fluticasone Furoate 55 µg Per Day | Placebo
Number analyzed (Participants) | 131 | 130
Scores on a scale
  Entire Treatment Period, n=131, 130 | -0.46 (0.09) | -0.32 (0.09)
  Week 1, n=131, 130 | -0.31 (0.09) | -0.22 (0.09)
  Week 2, n= 131, 128 | -0.61 (0.10) | -0.39 (0.10)

9. Secondary Outcome: Mean Change From Baseline (BL) in the Total Ocular Symptom Score (TOSS) for the Baseline TOSS >0 Over the Entire Treatment Period, at Week 1, and at Week 2
Description: as for outcome 8
Time Frame: Baseline through the entire treatment period (2 weeks), Week 1, and Week 2
Population: FAS. Only those participants with BL TOSS >0 who were available for assessment at both BL and the indicated assessment period were analyzed. Participants were analyzed for the entire treatment period if they had an assessment on any day during Week 1 and Week 2. Analysis was based on an ANCOVA with a model adjusting for Treatment, BL, Age, and Sex.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Fluticasone Furoate 55 µg Per Day | Placebo
Number analyzed (Participants) | 99 | 92
Scores on a scale
  Entire Treatment Period, n=99, 92 | -0.77 (0.11) | -0.47 (0.11)
  Week 1, n=99, 92 | -0.56 (0.11) | -0.35 (0.11)
  Week 2, n= 99, 90 | -0.99 (0.13) | -0.56 (0.13)

10. Secondary Outcome: Mean Percent Change From Baseline (BL) in the TOSS Over the Entire Treatment Period, at Week 1, and at Week 2
Description: Symptoms of eye itching, tearing, and redness were scored by the participant's (par.) parent/guardian who signed the ICF or the par. themself using a scale of 0, 1, 2, or 3 (a larger score indicates more severe symptoms) and were recorded in the par.'s diary. The TOSS is the sum of all 3 symptom scores and ranges from 0 to 9. The mean of the BL period is defined as the mean score of 4 consecutive days prior to Visit 2 (start of the treatment period). The mean of each assessment period is defined as the mean score of the entire treatment period (Weeks 1 and 2), Week 1, and Week 2. For each assessment period, a mean score for each par. was calculated using available diary data from the assessment periods, taking the average of non-missing data during the period. Percent change from BL=(mean score at post-BL assessment minus score at BL) divided by the BL value * 100. Par. with a BL TOSS of 0 were not analyzed because percent change from BL could not be calculated.
Time Frame: Baseline through the entire treatment period (2 weeks), Week 1, and Week 2
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Fluticasone Furoate 55 µg Per Day | Placebo
Number analyzed (Participants) | 99 | 92
Percent change
  Entire Treatment Period, n=99, 92 | -20.97 (11.39) | 1.57 (11.64)
  Week 1, n=99, 92 | -9.20 (10.90) | 5.37 (11.14)
  Week 2, n= 99, 90 | -33.52 (13.27) | -1.70 (13.69)

11. Secondary Outcome: Mean Percent Change From Baseline (BL) in the TOSS for the Baseline TOSS >0 Over the Entire Treatment Period, at Week 1, and at Week 2
Description: Symptoms of eye itching, tearing, and redness were scored by the participant's (par.) parent/guardian who signed the ICF or the par. themself using a scale of 0, 1, 2, or 3 (a larger score indicates more severe symptoms) and were recorded in the par.'s diary. The TOSS is the sum of all 3 symptom scores and ranges from 0 to 9. The mean of the BL period is defined as the mean score of 4 consecutive days prior to Visit 2 (start of the treatment period). The mean of each assessment period is defined as the mean score of the entire treatment period (Weeks 1 and 2), Week 1, and Week 2. For each assessment period, a mean score for each par. was calculated using available diary data from the assessment periods, taking the average of non-missing data during the period. Percent change from BL=(mean score at post-BL assessment minus score at BL) divided by the BL value * 100.
Time Frame: Baseline through the entire treatment period (2 weeks), Week 1, and Week 2
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Fluticasone Furoate 55 µg Per Day | Placebo
Number analyzed (Participants) | 99 | 92
Percent change
  Entire Treatment Period, n=99, 92 | -20.97 (11.39) | 1.57 (11.64)
  Week 1, n=99, 92 | -9.20 (10.90) | 5.37 (11.14)
  Week 2, n=99, 90 | -33.52 (13.27) | -1.70 (13.69)

12. Secondary Outcome: Mean Change From Baseline in the Individual Ocular Symptom Scores (Eye Itching, Tearing, and Redness) Over the Entire Treatment Period, at Week 1, and at Week 2
Description: Symptoms of eye itching, tearing, and redness were scored by the participant's parent/guardian who signed the ICF or the participant themself using a scale of 0, 1, 2, or 3 (a larger score indicates more severe symptoms) and were recorded in the participant's diary. The mean of the Baseline period is defined as the mean score of 4 consecutive days prior to Visit 2 (start of the treatment period). The mean of each assessment period is defined as the mean score of the entire treatment period (Weeks 1 and 2), Week 1, and Week 2. For each assessment period, a mean score for each participant was calculated using available diary data from the assessment periods, taking the average of non-missing data during the period. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline through the entire treatment period (2 weeks), Week 1, and Week 2
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Fluticasone Furoate 55 µg Per Day | Placebo
Number analyzed (Participants) | 131 | 130
Scores on a scale
  Eye itching, Entire Treatment Period, n=131, 130 | -0.24 (0.04) | -0.18 (0.04)
  Eye itching, Week 1, n=131, 130 | -0.15 (0.04) | -0.13 (0.04)
  Eye itching Week 2, n=131, 128 | -0.34 (0.05) | -0.23 (0.05)
  Tearing, Entire Treatment Period, n=131, 130 | -0.10 (0.03) | -0.05 (0.03)
  Tearing, Week 1, n=131, 130 | -0.09 (0.03) | -0.03 (0.03)
  Tearing, Week 2, n=131, 128 | -0.11 (0.03) | -0.07 (0.03)
  Redness, Entire Treatment Period, n=131, 130 | -0.11 (0.03) | -0.09 (0.03)
  Redness, Week 1, n=131, 130 | -0.07 (0.03) | -0.07 (0.03)
  Redness, Week 2, n=130, 128 | -0.16 (0.04) | -0.10 (0.04)

13. Secondary Outcome: Mean Change From Baseline in the Score of Troubles With Daily Life Over the Entire Treatment Period, at Week 1, and at Week 2
Description: The participant's parent/guardian who signed the ICF or the participant themself scored the participant's troubles with daily life once daily using the following scale: 0, None; 1, Few troubles; 2, Intermediate between 3 and 1; or 3, Painful and complicating daily life. The mean of the Baseline period is defined as the mean score of 4 consecutive days prior to Visit 2 (start of the treatment period). The mean of each assessment period is defined as the mean score of the entire treatment period (Weeks 1 and 2), Week 1, and Week 2. For each assessment period, a mean score for each participant was calculated using available diary data from the assessment periods, taking the average of non-missing data during the period. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline through the entire treatment period (2 weeks), Week 1, and Week 2
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Fluticasone Furoate 55 µg Per Day | Placebo
Number analyzed (Participants) | 131 | 130
Scores on a scale
  Entire Treatment Period, n=131, 130 | -0.43 (0.04) | -0.13 (0.04)
  Week 1, n=131, 130 | -0.33 (0.04) | -0.10 (0.04)
  Week 2, n=131, 128 | -0.53 (0.05) | -0.16 (0.05)

14. Secondary Outcome: Number of Participants With the Indicated Scores for Rhinoscopy Findings (Swelling of Inferior Turbinate Mucosa, Color of Inferior Turbinate Mucosa, Quantity of Nasal Discharge, and Quality of Nasal Discharge) at Baseline, Week 1, and Week 2/EW
Description: Rhinoscopy was assessed by the investigator by scoring swelling of inferior turbinate mucosa (SOITM) scored as 0 (none), 1 (possible to see center of the middle turbinate), 2 (between 3 and 1), or 3 (impossible to see middle turbinate); color of inferior turbinate mucosa (COITM) scored as 0 (normal), 1 (pink), 2 (red), or 3 (pale); quantity of nasal discharge (QTND) scored as 0 (none), 1 (small amount adhered), 2 (between 3 and 1), or 3 (filled); and quality of nasal discharge (QLND) scored as 0 (none), 1 (pyoid), 2 (viscous), or 3 (watery).
Time Frame: Baseline, Week 1, and Week 2/Early Withdrawal (EW)
Population: FAS. Participants who were withdrawn before Visit 3 (Week 1) were not included in the analysis for Week 1.
Measure: Number; unit: participants
Arm/Group | Fluticasone Furoate 55 µg Per Day | Placebo
Number analyzed (Participants) | 131 | 130
participants
  SOITM, Baseline, Score 0, n=131, 130 | 2 | 7
  SOITM, Baseline, Score 1, n=131, 130 | 24 | 32
  SOITM, Baseline, Score 2, n=131, 130 | 54 | 55
  SOITM, Baseline, Score 3, n=131, 130 | 51 | 36
  SOITM, Week 1, Score 0, n=131, 128 | 9 | 5
  SOITM, Week 1, Score 1, n=131, 128 | 45 | 55
  SOITM, Week 1, Score 2, n=131, 128 | 53 | 44
  SOITM, Week 1, Score 3, n=131, 128 | 24 | 24
  SOITM, Week 2/EW, Score 0, n=131, 130 | 19 | 19
  SOITM, Week 2/EW, Score 1, n=131, 130 | 62 | 45
  SOITM, Week 2/EW, Score 2, n=131, 130 | 37 | 42
  SOITM, Week 2/EW, Score 3, n=131, 130 | 13 | 24
  COITM, Baseline, Score 0, n=131, 130 | 2 | 2
  COITM, Baseline, Score 1, n=131, 130 | 13 | 31
  COITM, Baseline, Score 2, n=131, 130 | 28 | 29
  COITM, Baseline, Score 3, n=131, 130 | 88 | 68
  COITM, Week 1, Score 0, n= 131, 128 | 5 | 2
  COITM, Week 1, Score 1, n= 131, 128 | 45 | 43
  COITM, Week 1, Score 2, n= 131, 128 | 23 | 27
  COITM, Week 1, Score 3, n= 131, 128 | 58 | 56
  COITM, Week 2/EW, Score 0, n=131, 130 | 7 | 10
  COITM, Week 2/EW, Score 1, n=131, 130 | 68 | 51
  COITM, Week 2/EW, Score 2, n=131, 130 | 17 | 20
  COITM, Week 2/EW, Score 3, n=131, 130 | 39 | 49
  QTND, Baseline, Score 0, n=131, 130 | 8 | 6
  QTND, Baseline, Score 1, n=131, 130 | 52 | 53
  QTND, Baseline, Score 2, n=131, 130 | 60 | 63
  QTND, Baseline, Score 3, n=131, 130 | 11 | 8
  QTND, Week 1, Score 0, n= 131, 128 | 38 | 18
  QTND, Week 1, Score 1, n= 131, 128 | 57 | 62
  QTND, Week 1, Score 2, n= 131, 128 | 32 | 42
  QTND, Week 1, Score 3, n= 131, 128 | 4 | 6
  QTND, Week 2/EW, Score 0, n=131, 130 | 63 | 37
  QTND, Week 2/EW, Score 1, n=131, 130 | 49 | 57
  QTND, Week 2/EW, Score 2, n=131, 130 | 18 | 31
  QTND, Week 2/EW, Score 3, n=131, 130 | 1 | 5
  QLND, Baseline, Score 0, n=131, 130 | 9 | 6
  QLND, Baseline, Score 1, n=131, 130 | 0 | 0
  QLND, Baseline, Score 2, n=131, 130 | 29 | 27
  QLND, Baseline, Score 3, n=131, 130 | 93 | 97
  QLND, Week 1, Score 0, n= 131, 128 | 39 | 18
  QLND, Week 1, Score 1, n= 131, 128 | 2 | 5
  QLND, Week 1, Score 2, n= 131, 128 | 24 | 27
  QLND, Week 1, Score 3, n= 131, 128 | 66 | 78
  QLND, Week 2/EW, Score 0, n=131, 130 | 62 | 33
  QLND, Week 2/EW, Score 1, n=131, 130 | 3 | 3
  QLND, Week 2/EW, Score 2, n=131, 130 | 26 | 29
  QLND, Week 2/EW, Score 3, n=131, 130 | 40 | 65

15. Secondary Outcome: Number of Participants With the Indicated Overall Response to Therapy, as Assessed by the Investigator
Description: The investigator evaluated the participant's overall response to therapy (defined as improvement in the symptoms of allergic rhinitis) compared with Visit 2 (start of the treatment period), using the following 7-point categorical scale: 1=significantly improved, 2=moderately improved, 3=mildly improved, 4=no change, 5=mildly worse, 6=moderately worse, and 7=significantly worse.
Time Frame: Week 2/EW
Population: FAS
Measure: Number; unit: participants
Arm/Group | Fluticasone Furoate 55 µg Per Day | Placebo
Number analyzed (Participants) | 131 | 130
participants
  Significantly improved | 32 | 12
  Moderately improved | 38 | 25
  Mildly improved | 36 | 31
  No change | 22 | 54
  Mildly worse | 1 | 5
  Moderately worse | 2 | 2
  Significantly worse | 0 | 1

16. Secondary Outcome: Number of Participants With the Indicated Overall Response to Therapy, as Assessed by the Participant's Parent/Guardian or the Participant
Description: The participant's parent/guardian who signed the ICF or the participant themself evaluated the participant's overall response to therapy (defined as improvement in the symptoms of allergic rhinitis) compared with Visit 2 (start of the treatment period), using the following 7-point categorical scale: 1=significantly improved, 2=moderately improved, 3=mildly improved, 4=no change, 5=mildly worse, 6=moderately worse, and 7=significantly worse.
Time Frame: Week 2/EW
Population: FAS
Measure: Number; unit: participants
Arm/Group | Fluticasone Furoate 55 µg Per Day | Placebo
Number analyzed (Participants) | 131 | 130
participants
  Significantly improved | 28 | 2
  Moderately improved | 51 | 26
  Mildly improved | 34 | 48
  No change | 18 | 51
  Mildly worse | 0 | 3
  Moderately worse | 0 | 0
  Significantly worse | 0 | 0

ADVERSE EVENTS:
Time Frame: Participants were analyzed from the start of study treatment until the follow up contact (up to 3 weeks).
Description: Serious adverse events (SAEs) and non-serious adverse events (AEs) were collected in the Safety Population, comprised of all randomized participants who received at least one dose of study medication, according to the actual treatment received.
Arm/Group | Fluticasone Furoate 55 µg Per Day | Placebo
Serious Adverse Events (participants affected / at risk) | 0/131 | 0/130
Other Adverse Events (participants affected / at risk) | 23/131 | 25/130
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluticasone Furoate 55 µg Per Day (N=131) | Placebo (N=130)
Nasopharyngitis (Infections and infestations) | 6 | 3
Bronchitis (Infections and infestations) | 1 | 1
Acute sinusitis (Infections and infestations) | 1 | 0
Conjunctivitis bacterial (Infections and infestations) | 1 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 1 | 0
Impetigo (Infections and infestations) | 1 | 0
Otitis media acute (Infections and infestations) | 0 | 1
Pneumonia mycoplasmal (Infections and infestations) | 0 | 1
Streptococcal infection (Infections and infestations) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Heat illness (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 2
Blood potassium increased (Investigations) | 0 | 1
Eosinophil count increased (Investigations) | 1 | 0
Conjunctivitis allergic (Eye disorders) | 2 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 2
Orthostatic intolerance (Nervous system disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Heat rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 1
Ear discomfort (Ear and labyrinth disorders) | 1 | 0
Tooth extraction (Surgical and medical procedures) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.